CLINICAL TRIAL: NCT05491759
Title: A Randomised Three-way Cross Over Study to Determine the Optimal Absorption of an Omega-3 Supplement Administered as a Single Oral Dose to Healthy Volunteers
Brief Title: A Study to Determine Optimal Absorption of Single Dose Omega-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: BTFISH-22
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2022-12

CONDITIONS: Optimal Gastrointestinal Absorption of Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Product 1 - AquaCelle Fish Oil Triglyceride (Experimental): 1 dose of 2 capsules equivalent to 1.6g Fish Oil Triglyceride (standardised to contain 1120 mg of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA)) and 0.4g AquaCelle The dose will be consumed orally with 250 mL water.
  Interventions: Drug: Product 1 - AquaCelle Fish Oil Triglyceride
- Product 2 - AquaCelle Fish Oil Ethyl Ester (Experimental): 1 dose of 2 capsules equivalent to 1.6g Fish Oil Ethyl Ester (standardised to contain 1120 mg of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA)) and 0.28g AquaCelle The dose will be consumed orally with 250 mL water.
  Interventions: Drug: Product 2 - AquaCelle Fish Oil Ethyl Ester
- Product 3 - Standard Fish Oil Triglyceride (Experimental): 1 dose of 2 capsules equivalent to 1.6g Fish Oil Triglyceride (standardised to contain 1120 mg of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA)).
  The dose will be consumed orally with 250 mL water.
  Interventions: Drug: Product 3 - Standard Fish Oil Triglyceride

INTERVENTIONS:
Drug: Product 1 - AquaCelle Fish Oil Triglyceride — 1 dose of 2 capsules equivalent to 1.6g Fish Oil Triglyceride (standardised to contain 1120 mg of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA)) and 0.4g AquaCelle.
  Arms: Product 1 - AquaCelle Fish Oil Triglyceride
Drug: Product 2 - AquaCelle Fish Oil Ethyl Ester — 1 dose of 2 capsules equivalent to 1.6g Fish Oil Ethyl Ester (standardised to contain 1120 mg of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA)) and 0.28g AquaCelle
  Arms: Product 2 - AquaCelle Fish Oil Ethyl Ester
Drug: Product 3 - Standard Fish Oil Triglyceride — 1 dose of 2 capsules equivalent to 1.6g Fish Oil Triglyceride (standardised to contain 1120 mg of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA)).
  Arms: Product 3 - Standard Fish Oil Triglyceride

SUMMARY:
This is a randomised three-way cross over study comparing the optimal absorption of a single dose of fish oil using 3 different forms to one another on increasing blood concentrations of fatty acids in 24 healthy adult participants aged 19 years and over.

ELIGIBILITY:
Inclusion Criteria:

* Male and females over 19 years and otherwise healthy
* Healthy BMI >18.0 and <30.0
* Able to provide informed consent
* Agree to arrive fasted on the day of the trial
* Agree to participate in all arms of the study

Exclusion Criteria:

* Unstable or serious illness [e.g. kidney, liver (including NAFLD), GIT, heart conditions, diabetes, thyroid gland function malignancy]*
* Any treatment that included radiation or chemotherapy within the previous 2 years
* Receiving/prescribed coumandin (Warfarin), heparin, daltaparin, enoxaparin or other anticoagulation therapy.
* Regular use of supplements containing the investigational material (e.g. Omega-3 fatty acids), in the last 3 months, regular consumption of foods containing the investigational material (e.g. fish for omega-3) #
* Active smokers, nicotine, alcohol, drug abuse
* Chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Allergic to any of the ingredients (i.e., fish oil)
* Pregnant or lactating women
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion

  * An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

    * Regular use or consumption is considered if participants are consuming omega containing supplements or foods on 3 or more days per week.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Plasma EPA+DHA as measured by AUC0-24 | 0, 2, 4, 6, 8, 10, 12 and 24 hours post ingestion
  Change in plasma EPA+DHA from baseline as measured by AUC0-24

SECONDARY OUTCOMES:
Cmax | 24 hours post ingestion
  Peak plasma concentration
Tmax | 24 hours post ingestion
  Time to peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: David Briskey, PhD, Principal Investigator — The University of Queensland
Locations (1):
- RDC Global Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared